CLINICAL TRIAL: NCT00968500
Title: Understanding the Psychosocial Needs of Parents Who Have Lost a Child to Cancer
Status: Active, not recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Dana-Farber Cancer Institute (Other); Ohio State University (Other); University of Memphis (Other); University of Southern California (Other)
Responsible Party: Sponsor
Other Study IDs: 09-107; NCT01324154 (obsolete NCT alias)
Record Dates: First submitted 2009-08-28; First posted 2009-08-31 (Estimated); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Parents Who Have Lost a Child to Cancer
Keywords: Grief; bereavement; questionnaires; 09-107
MeSH Terms: interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Parents Who Have Lost a Child to Cancer: The overall goal of the proposed cross-sectional study is to obtain information necessary to the development of an effective Meaning-Centered Grief Intervention for parents who lost a child to cancer. In order to identify a subset of parents with whom we will conduct qualitative interviews with a subset of participants to address Aims 1 and 2, we will first screen participants to determine their levels of Prolonged Grief Disorder symptoms using a quantitative assessment (PG-13). The screening measure (PG-13) and the additional questionnaires included in the quantitative battery of measures will be analyzed to achieve Aim 3.
  Interventions: Behavioral: Questionnaires/Interviews

INTERVENTIONS:
Behavioral: Questionnaires/Interviews — Prior to the interview, the measure of prolonged grief disorder symptoms, the PG-13, will be re-administered to participants as a quality assurance check. We will administer 7 self-report measures, which participants can complete in our office, at home, or via telephone, depending on their preferences. These questionnaires should take approximately 75 to 80 minutes to complete. If you are asked to take part in the in-depth interview and you choose to take part, the interview that will take approximately 60 to 90 minutes to complete, depending on the length of the responses to the questions asked.
  The participant may also be asked if they would be willing to fill out an additional questionnaire about parents' thoughts on the most appropriate timing for raising the topic of a postmortem examination and factors that are important to include in discussions. Despite its importance, autopsy is often not discussed with parents whose child is dying from cancer.

SUMMARY:
The purpose of this study is to understand the experiences and needs of parents who have lost a child to cancer. This will aid us in developing an intervention that may help parents cope with their loss.

ELIGIBILITY:
Inclusion Criteria:

* Loss of a child to cancer between 6 months and 6 years ago
* Loss of a child between the ages of 6 months and 25 years
* Biological or adoptive parent or stepparent
* Parent must be age 18 or over
* In the judgment of investigators/consenting professionals able to comprehend English to complete study assessments
* To be eligible for the qualitative interview, participants more score of 19 or less (< 19)or 34 or greater (> 34) on the PG-13 to qualify

Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator's judgment, to preclude completion of the assessment measures, interview or informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Bereaved parents will be identified through death records kept by the Department of Pediatrics and cross-referenced with the deceased child's MSK medical record.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2009-08; Primary Completion 2027-06-02 (Estimated); Study Completion 2027-06-02 (Estimated)

PRIMARY OUTCOMES:
Identify the unique qualitative themes related to finding meaning among parents who lost a child to cancer to inform development of a conceptually sound meaning-centered grief intervention. | 2 years

SECONDARY OUTCOMES:
Determine differences in qualitative themes of meaning in parents in the high and low Prolonged Grief Disorder subgroups to help select a target population for a meaning-centered grief intervention. | 2 years
Explore and identify factors associated with bereaved parents' psychosocial service underutilization to guide the development of an acceptable and feasible meaning-centered grief intervention format. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian Nelson, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - NCI Clinical Center, Bethesda, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm